CLINICAL TRIAL: NCT01490892
Title: Quantitative Subharmonic Breast Imaging
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Lantheus Medical Imaging (Industry); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11F.438; R01CA140338 (NIH); JT 2179 (Other: JeffTrial Number)
Record Dates: First submitted 2011-12-08; First posted 2011-12-13 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: breast abnormality; ultrasound imaging; ultrasound contrast agent; subharmonic imaging
MeSH Terms: conditions — Breast Neoplasms | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3D HI and SHI of UCA (Experimental): Perflutren injection, suspension (IV)0.25 ml followed by 3D Harmonic imaging (HI) then (IV) 20 micro-l/kg followed by 3D subharmonic imaging (SHI)
  Interventions: Drug: 3D HI and SHI of UCA

INTERVENTIONS:
Drug: 3D HI and SHI of UCA — Perflutren injection, suspension (IV)0.25 ml followed by 3D Harmonic imaging (HI) then (IV) 20 micro-l/kg followed by 3D subharmonic imaging (SHI)
  Other Names: Definity

SUMMARY:
This is a non-randomized trial of 450 women with a breast abnormality, who are scheduled for a breast biopsy of this abnormality. The study will be conducted at two clinical sites. The primary objective of this trial is:

To evaluate if quantitative 3D Subharmonic imaging (SHI) or pulse inversion harmonic imaging (HI) can improve the characterization of benign and malignant breast masses (independently or in combination with other imaging modes) compared to x-ray mammography, fundamental grayscale ultrasound (US) or power Doppler imaging (PDI).

The secondary aim of this trial is:

To compare quantitative (bifurcations & vessel length) and semi-quantitative (blood pool & parametric imaging) measures of the vascular morphology of breast lesions determined by pathology and by SHI.

DETAILED DESCRIPTION:
This is an open-label, non-randomized trial that will be conducted at two clinical sites (the Breast Imaging Centers at Thomas Jefferson University (TJU) Hospital and University of California, San Diego (UCSD) Hospital). All 450 subjects will receive at most two IV bolus injections of Definity (Lantheus Medical Imaging, Billerica, MA), will undergo an unenhanced (baseline) and Definity contrast-enhanced US imaging study for evaluation of a breast mass or breast abnormality without mass, and will be scheduled to undergo a clinically indicated biopsy of the breast lesion under investigation.

ELIGIBILITY:
Inclusion Criteria:

* Be a female diagnosed by x-ray mammography (performed within 90 days prior to the study procedure) as having a solid breast mass or abnormal area without a mass.
* Be scheduled for a biopsy (core / excisional / lumpectomy) of the mass or region of abnormality or for mastectomy within 30 days after this study procedure.
* Be at least 18 years of age.
* Be medically stable.
* If a female of child-bearing potential, must have a negative pregnancy test.
* Have signed Informed Consent to participate in the study.

Exclusion Criteria:

* Males
* Females who are pregnant or nursing.
* Patients whose breast lesion is unequivocally a cyst by unenhanced US.
* Patients currently on chemotherapy or with other primary cancers requiring systemic treatment.
* Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable. For example:
* Patients on life support or in a critical care unit.
* Patients with unstable occlusive disease (eg, crescendo angina)
* Patients with clinically unstable cardiac arrhythmias, such as recurrent ventricular tachycardia.
* Patients with uncontrolled congestive heart failure (NYHA Class IV)
* Patients with recent cerebral hemorrhage.
* Patients with clinically significant and unstable renal and/or liver disease (eg, transplant recipients in rejection)
* Patients who have undergone surgery within 24 hours prior to the study sonographic examination.
* Patients with known hypersensitivity to perflutren
* Patients who have received any contrast medium (X-ray, MRI, CT, of US) in the 24 hours prior to the research US exam
* Patients with cardiac shunts.
* Patients with congenital heart defects.
* Patients with severe emphysema, pulmonary vasculitis, or a history of pulmonary emboli.
* Patients with confirmed or suspected liver lesions.
* Patients with respiratory distress syndrome.
* Patients who have had excisional biopsy/lumpectomy of the current area of interest within the past 6 weeks.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2011-11; Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Forsberg, phD, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - University of California, San Diego, La Jolla, California
  - Thomas Jefferson University, Dept of Radiology, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Forsberg F, Piccoli CW, Merton DA, Palazzo JJ, Hall AL. Breast lesions: imaging with contrast-enhanced subharmonic US--initial experience. Radiology. 2007 Sep;244(3):718-26. doi: 10.1148/radiol.2443061588. Epub 2007 Aug 9. PMID 17690324

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3D HI and SHI of UCA
Started | 219
Completed | 219
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 3D HI and SHI of UCA
Number analyzed (Participants) | 219
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 175
  >=65 years | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 219
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 204
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 97
  White | 108
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 219

OUTCOME MEASURES:

1. Primary Outcome: Number of Breast Cancer Lesions Characterized as Malignant or Benign With 3D SHI, Harmonic Imaging (HI) or Power Doppler Imaging (PDI)
Description: Characterization of benign and malignant breast cancer lesions is compared by each imaging method which evaluates vascular activity. Imaging methods to be compared are 3D Subharmonic imaging (SHI) or pulse inversion harmonic imaging (HI), fundamental grayscale ultrasound (US) or power Doppler imaging (PDI). Data will be analyzed qualitatively.
Time Frame: 2 hours
Measure: Number; unit: lesions
Arm/Group | 3D HI and SHI of UCA
Number analyzed (Participants) | 219
lesions
  Power Doppler Imaging (PDI) : Benign | 69
  Power Doppler Imaging (PDI) : Malignant | 24
  Power Doppler Imaging (PDI) : Not Characterized | 126
  3D SHI : Benign | 58
  3D SHI : Malignant | 25
  3D SHI : Not Characterized | 136
  Harmonic Imaging (HI) : Benign | 3
  Harmonic Imaging (HI) : Malignant | 5
  Harmonic Imaging (HI) : Not Characterized | 211

2. Secondary Outcome: Change in Vascular Volume of Breast Lesions as Assessed by Subharmonic Imaging (SHI) Signal Intensity
Description: Quantitative measures of the vascular volumes of breast lesions determined by SHI utilizing bifurcations and vessel length, and blood pool and parametric imaging
Time Frame: 2 hours
Population: breast cancer lesions
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | 3D HI and SHI of UCA
Number analyzed (Participants) | 219
dB
  Central Benign lesions | 1.83 (0.16)
  Peripheral benign lesions | 1.5 (0.09)
  Central malignant lesions | 1.72 (0.33)
  peripheral malignant lesions | 1.26 (0.21)

ADVERSE EVENTS:
Time Frame: baseline to 30 minutes post contrast injection for Adverse Events, All-Cause Mortality up to 1 year
Arm/Group | 3D HI and SHI of UCA
All-Cause Mortality (participants affected / at risk) | 2/219
Serious Adverse Events (participants affected / at risk) | 0/219
Other Adverse Events (participants affected / at risk) | 0/219

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-07-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT01490892/Prot_SAP_000.pdf